CLINICAL TRIAL: NCT00499057
Title: Interstitial High Dose-Rate Brachytherapy for Partial Breast Irradiation in Early Breast Cancer: Results of Phase II Prospective Study
Brief Title: Partial Breast Irradiation With Interstitial High Dose Rate Brachytherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Cynthia Aristei, Full Professor of Rdaiotherapy, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRT-HDR
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
Keywords: early stage breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Other): single arm study
  Interventions: Radiation: interstitial high dose-rate brachytherapy, PBI

INTERVENTIONS:
Radiation: interstitial high dose-rate brachytherapy, PBI — Single arm study Treatment schedule is 4 Gy twice a day, with a time relapse of at least 6 hours between each fraction, for four days, for a total dose 32 Gy.

SUMMARY:
Partial breast irradiation (PBI) is becoming more widespread in the treatment of early breast cancer in patients at low risk of relapse as pathological and clinical findings have demonstrated that most breast cancer recurrences after BCS occur close to the tumour bed. In our phase II prospective study PBI is administered with high-dose-rate brachytherapy in patients with low-risk early-stage breast cancer. Patients receive 4 Gy twice a day for 4 days (total dose 32 Gy).

DETAILED DESCRIPTION:
Patients included in our phase II trial of PBI with interstitial HDR brachytherapy are at low-risk of relapse. Implants are positioned during surgery or postoperatively, within 12 weeks. Treatment schedule is 4 Gy twice a day, with a time relapse of at least 6 hours between each fraction, for four days, for a total dose 32 Gy. Before post-operative implantation, all patients undergo a breast computed tomography (CT) scan to visualize and expand the excision cavity and obtain the planning target volume (PTV), i.e. the lumpectomy cavity plus a margin of 1-2 cm around it. Through virtual simulation with a 3D treatment planning system (TPS), we define the implant catheter position. After implantation, in all patients a breast CT scan checked implant geometry. On CT images transferred to a TPS the surgical cavity is outlined and expanded, the PTV defined, and inactive and active source lengths measured.CT-based 3D software is used to identify and reconstruct the catheters, outline and expand the surgical cavity and obtain the PTV. Dwell positions are activated for each catheter, and inactive and active lengths defined.Prescribed dose was 85% of the basal dose. Dwell weights are optimised in the basal points applying the volume and distance method and best values were chosen independently of strategy. A dose-volume histogram that records the volume covered by 100% and 150% of the prescribed dose (V100 and V150) was obtained for each patient. DHI, defined as V150 - V100/ V100 (7), is recognized as the most suitable quality index.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 40 years
* ECOG performance status 0-2
* T dimensions ≤ 2.5 cm
* Negative surgical margins
* Negative axillary lymph nodes
* Suitable breast anatomy for implantation

Exclusion Criteria:

* Age < 40 years
* ECOG performance status > 2
* T dimensions > 2.5
* Positive surgical margins
* Positive axillary lymph node
* Infiltrating lobular histology
* Significant areas of lobular carcinoma in situ
* Paget's disease of the nipple
* Extensive intraductal component (EIC)
* Lymphovascular invasion
* Multifocality (n) skin infiltration

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-08; Primary Completion 2015-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
cancer related deaths | 6 months
local relapses | 6 months

SECONDARY OUTCOMES:
quality of life | 6 months
cosmetic results | 6 months
toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Aristei, Prof. M.D., Study Director — University Of Perugia
Locations (1):
- Radiation Oncology Institute, Perugia, Perugia, Italy

REFERENCES:
- [Derived] Aristei C, Palumbo I, Capezzali G, Farneti A, Bini V, Falcinelli L, Margaritelli M, Lancellotta V, Zucchetti C, Perrucci E. Outcome of a phase II prospective study on partial breast irradiation with interstitial multi-catheter high-dose-rate brachytherapy. Radiother Oncol. 2013 Aug;108(2):236-41. doi: 10.1016/j.radonc.2013.08.005. Epub 2013 Sep 14. PMID 24044802